CLINICAL TRIAL: NCT02420600
Title: The Clinical Relevance of Immune Cells and Circulating Tumor Cells in Patients With Head and Neck Cancer
Brief Title: The Clinical Relevance of Immune Cells and CTC in HNSCC Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CTCHNSCC02; CMRPG3E0511-0512 (Other: Grantor or Funder CMRPG3E0511-0512)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-04

CONDITIONS: Recurrence; Metastasis; Death
Keywords: Circulating tumor cells; Head and neck cancer; PD-1; natural killer cells; cytotoxic T lymphocytes
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis; Death; Neoplastic Cells, Circulating; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Head and neck squamous cell carcinomas (HNSCCs) are mainly caused by tobacco, alcohol consumption and betel nut chewing and the sixth most common cancer in the world. Despite significant advances in the treatment modalities involving surgery, radiotherapy, and concomitant chemoradiotherapy, the 5-year survival rate remained below 50% for the past 30 years.

The worse prognosis of these cancers must certainly be linked to the fact that HNSCCs strongly influence the host immune system. During this process, mesenchymal tumor-like cells are highly mobile and enter quickly adjacent structure (intravasation), from where they travel through lymphatic and blood vessels as circulating tumor cells (CTC), which are single cells with malignant potential detected in the peripheral bloodstream and essential for establishing metastasis.

Programmed death 1 (PD-1) and its ligand (PD-L1) play pivotal roles in regulating host immune responses. Substantial evidence has demonstrated that PD-L1 can deliver an inhibitory signal to PD-1 expressing T cells, leading to suppression of the immune response by inducing apoptosis, energy, unresponsiveness and functional exhaustion of T cells. However, the inhibitory effects of this pathway on the function of cytotoxic T lymphocytes, the main effector cells in HNSCC patients, are not well defined.

In this study aims to solve two main problems: one is to improve and try to optimize current protocols of CTC isolations based on the investigator previous work, which is one of most challenging problems in CTC field to date; the other is to understand the status of immune system in HNSCC patients, especially focusing on PD-1-PD-L1 pathway and its expressions. After series basic experiments of immune cell analysis and conditional adjustment of CTC isolation protocols, the investigator are willing to isolate CTCs and immune cells at a single blood drawing at the same time. A prospective trial will be conducted to elucidate the roles of PD-1 expression lymphocytes and CTC numbers on the clinical outcomes of HNSCC patients.

DETAILED DESCRIPTION:
1. To establish a platform to increase the efficiency and purity for isolation and enumeration of circulating tumor cells from patients with head and neck cancer.
2. Compare the differences and determine the most efficient method or combination of negative, positive selection, optoelectronic dielectrophoresis (ODEP) and flow cytometry sorting technology.

   1. Negative Selection
   2. Positive Selection
   3. ODEP devices
   4. Flow Cytometry and Sorting System
3. Use the upgraded platform and test among different groups for efficiency test. (Planned subjects: healthy donor: n=30; early-stage (stage I=II) patients=9; locally-advanced=9 and metastatic, n=9; total n=60)

   - Clinical Enrollment for Device/Method Validation
4. To confirm programmed death-1(PD-1) expression could be successfully detected and up-regulated on cytotoxic T cells using cell lines natural killer cell (NK-92).

   1. Cell Culture of NK-92, OECM-1, SCC-4 and K562
   2. Immunostaining methods for PD-1 expression
   3. Flow cytometry for ratio of PD-1 expression
5. To observe the functional changes of the cytotoxic T cells with PD-1 expression using cell lines and immunomagnetic bead-based isolation method.

   1. Positive Isolation for PD-1 Expressing Cells
   2. CD107a cytotoxicity assay
   3. Cell-mediated cytotoxicity assays
6. Confirm these findings in whole blood sample from healthy donors (n=15) and HNSCC patients (n=15).

   - Clinical Enrollment Patients for PD-1 expression in PBMCs, a stage of validation previous findings
7. Using the platform established on first-year project, to isolate and check the CTC number from locally advanced or metastatic HNSCC patients for validation.
8. To check the ratio of circulating CD56+ cells with PD-1 expression from locally advanced or metastatic HNSCC patients for validation.
9. To correlate the clinical relevance of circulating PD-1+CD56 cells and CTCs in locally advanced or metastatic HNSCC patients (N=60 in this year). Another Healthy donors (n=15) will be needed for reference.

   1. CTC enumeration and sorting technique-Negative Selection Strategy
   2. Positive Selection
   3. ODEP devices
   4. Flow Cytometry and Sorting System
   5. Clinical Enrollment HNSCC Patients for CTCs and PD-1 ratio

ELIGIBILITY:
Inclusion Criteria:

1. Established head and neck squamous cell carcinoma.
2. Age >=20 years old with clear consciousness, decided by free wills.

Ability to sign informed consent

Exclusion Criteria:

1. Patient's refusal
2. Poor compliance, cannot draw blood for CTCs isolation as time schedule or clinical treatment or follow-up
3. Difficult blood sampling
4. No more needs for CTCs evaluation, decided by clinicians.

Inability to comply with study and/or follow-up procedures.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Locally advanced or recurrent/metastatic head and neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The correlation among CTC numbers, PD-1 expressions and the prognosis of patients. | one year
  The CTCs will be isolated and then the number of CTCs will be measured. PD-1 expression from locally advanced or metastatic HNSCC patients will be validated. Measure response or progression events via all available imaging studies, including Chest-Xray, CT scans, or MRI, PET study. The relationship between CTCs number, PD1 expression and time from CTCs checkpoint to disease progression will be analyzed.

SECONDARY OUTCOMES:
Overall survival | one year
  All causes of death would be documented and the relationship between CTCs number and time from CTCs checkpoint to death will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsun Hsieh, M.D, M.S., Principal Investigator — Division of Hematology-Oncology, Department of Internal Medicine, Chang Gung Memorial Hospital at Lingkou
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Result] Hsieh JC, Lin HC, Huang CY, Hsu HL, Wu TM, Lee CL, Chen MC, Wang HM, Tseng CP. Prognostic value of circulating tumor cells with podoplanin expression in patients with locally advanced or metastatic head and neck squamous cell carcinoma. Head Neck. 2015 Oct;37(10):1448-55. doi: 10.1002/hed.23779. Epub 2014 Jul 24. PMID 24844673
- [Derived] Chang PH, Wu MH, Liu SY, Wang HM, Huang WK, Liao CT, Yen TC, Ng SH, Chen JS, Lin YC, Lin HC, Hsieh JC. The Prognostic Roles of Pretreatment Circulating Tumor Cells, Circulating Cancer Stem-Like Cells, and Programmed Cell Death-1 Expression on Peripheral Lymphocytes in Patients with Initially Unresectable, Recurrent or Metastatic Head and Neck Cancer: An Exploratory Study of Three Biomarkers in One-time Blood Drawing. Cancers (Basel). 2019 Apr 15;11(4):540. doi: 10.3390/cancers11040540. PMID 30991692